CLINICAL TRIAL: NCT02478502
Title: Phase 2 Study Cabazitaxel as Salvage Treatment for Cisplatin-resistant Germ Cell
Brief Title: Testis CAB: Cabazitaxel as Salvage Treatment for Cisplatin-resistant Germ Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University Hospital, Akershus (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jan Oldenburg, MD, PhD, Coordinating Investigator, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1627 b; 2012-004418-32 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2015-06-23 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Testicular Cancer
Keywords: testicular cancer; cisplatin resistancy
MeSH Terms: conditions — Testicular Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (single arm study) (Experimental): Cabazitaxel 25 mg/m2 each 3. week (no other drugs will be administered)
  Interventions: Drug: cabazitaxel

INTERVENTIONS:
Drug: cabazitaxel — cabazitaxel is given to patients with progressive testicular cancer after cisplatin-based chemotherapy
  Other Names: Jevtana

SUMMARY:
Germ cell tumors belong to the most chemosensitive malignancies. Paclitaxel in combination with ifosfamide and cisplatin (TIP) has become a common regimen for salvage treatment of germ cell cancer.

Cabazitaxel may overcome resistance to docetaxel and paclitaxel and might have clinical activity in patients with metastatic and progressive germ cell tumors.

DETAILED DESCRIPTION:
Patients with metastatic germ cell cancer and relapse after two or more courses of cisplatin-based chemotherapy or after high-dose chemotherapy have a poor prognosis and no curative options. Taxanes in various combinations unfold cytotoxic effects on germ cell tumors resistant to conventional doses of cisplatin. Paclitaxel in combination with ifosfamide and cisplatin (TIP) has become a common regimen for salvage treatment of germ cell cancer. In most patients, however, resistance to paclitaxel, as evidenced by progression occurs.Cabazitaxel has been developed to overcome resistance to docetaxel and paclitaxel. It has shown efficacy in patients progressing during docetaxel therapy in a large phase III trial (TROPIC) in patients with castration-resistant prostate cancer. Furthermore, chemotherapy resistance might be less likely to develop in patients receiving cabazitaxel as compared to other taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥ 18 years old
* Histologically verified metastatic germ cell cancer (GCC) of the testicle or extragonadal GCC originating from retroperitoneum or mediastinum
* Disease progression during cisplatin-based chemotherapy or Disease progression or relapse after high-dose chemotherapy or Disease progression or relapse after at least 2 different cisplatin-based regimens
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0-2
* Life expectancy ≥ 3 months
* At baseline adequate function of liver, kidneys and bone marrow:

·Neutrophils ≥ 1.5 x 109/L·

* Hemoglobin ≥ 9.0 g/dL
* Platelets ≥ 100 x 109/L
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Total Bilirubin ≤ 1.0 x ULN
* Serum glutamate oxaloacetate transaminase (SGOT/AST) ≤ 1.5 x ULN
* Serum glutamate pyruvate transaminase (SGPT/ALT) < 1.5 x ULN

Exclusion Criteria:

* Systemic antitumor treatment within 21 days before study entry
* Simultaneous radiotherapy to the only target lesion
* Patients unwilling or unable to comply with the protocol
* Patients with unstable angina pectoris, myocardial infarction ≤ 6 months prior to first study treatment, congestive heart failure New York Heart Association (NYHA) III-IV or serious uncontrolled cardiac arrhythmias
* Patients with an active or uncontrolled infection
* Patients who have a history of another primary malignancy and are off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer
* Patients who have undergone major surgery within 4 weeks prior to starting study drug (e.g. intra-thoracic, intra-abdominal, or intra-pelvic) or significant traumatic injury, or who have not recovered from the side effects of any of the above within 6 weeks
* Patients who have participated in another interventional clinical trial within 30 days before study entry
* Other serious medical conditions that could impair the ability of the patient to participate in the study
* Active infection requiring systemic antibiotic-, anti-viral-, or anti-fungal medication
* Neuropathy ≥Grade 2 Common Terminology Criteria for Adverse Events (CTCAE)
* Patient with reproductive potential not implementing accepted and effective method of contraception during the whole study period and up to 6 months after the last dose of cabazitaxel
* One or more of the following cabazitaxel-specific requirements:

  * History of severe hypersensitivity reaction (≥ Grade 3) to docetaxel
  * History of severe hypersensitivity reaction (≥ Grade 3) to polysorbate 80 containing drugs
  * Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4 (CYP3A4) (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix A and B)
  * Concurrent or planned treatment with Organic anion transporting polypeptide1B1 (OATP1B1) substrates e.g. statins, valsartan, repaglinide which have to be taken within 12 hours before cabazitaxel application and 3 hours after the end of infusion, refer table 9

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate | after 3 and 6 cycles of cabazitaxel (9 and 18 weeks, respectively) as change from baseline (radiologic evaluation before first cycle of cabazitaxel)
  Recist 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jan Oldenburg, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (4):
- Rigshospitalet, Copenhagen, Denmark
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T), Meldola, Italy
- Oslo University Hospital, Oslo, Norway
- University Hospital of Uppsala, Department of Oncology, Uppsala, Sweden